CLINICAL TRIAL: NCT02765542
Title: Developing Accessible mHealth Programs for Depression Management in Bolivia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, John Piette, VA Senior Research Career Scientist, Professor of Health Behavior and Health Education and of Internal Medicine, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: HUM00087937
Record Dates: First submitted 2015-03-04; First posted 2016-05-06 (Estimated); Last update posted 2016-05-06 (Estimated); Status verified 2016-05

CONDITIONS: Depression
Keywords: Depression; mHealth; Interactive Voice Response; Bolivia; Mental health
MeSH Terms: conditions — Depression; Psychological Well-Being

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Automated phone calls (Experimental): Automated disease assessment & self-care support phone calls for up to 12 weeks.
  Interventions: Other: Automated disease assessment & self-care support phone calls

INTERVENTIONS:
Other: Automated disease assessment & self-care support phone calls — Automated disease assessment & self-care support phone calls for up to 12 weeks.

SUMMARY:
The purpose of the study is to evaluate the feasibility and potential impact of an automated phone system in monitoring and improving self-care and health outcomes among patients with depression in Bolivia.

DETAILED DESCRIPTION:
All patients will receive a weekly 10-15 minute automated phone call to their cell phone for disease assessment and self-care support for up to 12 weeks. During enrollment, the research team will explain how to use the automated phone system. During patients' automated calls, they will be asked questions about their self-care relevant to their diagnosis, symptoms of depression, and medication adherence (if patients are prescribed an anti-depressant). Based on the patient's self-report, they will receive targeted suggestions for how to improve their self-management. At the end of each automated call, patients will hear the phone number of their clinic, which they can call for a health problem or to disenroll from the program. At the time of recruitment, if possible, an initial automated call will be sent to the patient's phone so that they can learn what to expect and have the chance to ask questions of the research associate who will be present.

In the event that the patient reports a health or self-care problem during their call (i.e., the patient reports rarely or never taking their medication), a report will automatically be generated and sent by email to the research team plus the patient's designated clinician so that follow-up can take place. The secure email address will be verified with each clinician, and be password protected.

The intervention will last up to 12 weeks, after which the patient will have a follow-up meeting with the research team and will complete a survey about the program. All follow-ups will take place either in person or over the phone.

ELIGIBILITY:
Inclusion Criteria:

* 21-80 years of age
* PHQ-8 score of 10 or higher

Exclusion Criteria:

* Have diagnoses indicating a six-month life expectancy
* Prior inpatient psychiatric treatment
* Patients with probable bipolar disorder or cognitive impairment as indicated on validated screeners

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2014-07; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Change from baseline on depressive symptoms at 12 weeks (PHQ-8 Scores) | Baseline and 12 week post-intervention follow-up

SECONDARY OUTCOMES:
Change from baseline on self-care behaviors at 12 weeks (self-care behavior questionnaire) | Baseline and 12 week post-intervention follow-up
Evaluate program feasibility (telephone call completion rates) | 12 week post-intervention follow-up
Patient satisfaction (satisfaction questionnaire) | 12 week Post-intervention follow-up
Patient qualitative feedback (qualitative questionnaire) | 12 week Post-intervention follow-up

CONTACTS AND LOCATIONS:
Overall Officials: John D Piette, PhD, Principal Investigator — University of Michigan
Locations (1):
- El Servicio Departmental de Salud (SEDES) affiliated clinics, La Paz, Bolivia

IPD SHARING:
Plan to Share IPD: No